CLINICAL TRIAL: NCT02883777
Title: Effect of a High Protein and Low Glycemic Index Diet on Kidney Transplant
Brief Title: Effect of a High Protein and Low Glycemic Index Diet on Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160121
Record Dates: First submitted 2016-08-03; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Failure, Chronic; End-Stage Renal Disease
Keywords: Kidney Transplantation; Low Glycemic Index; High Protein
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Protein and Low Glycemic Index Diet (Experimental): A protocol of a high protein and low glycemic index diet.
  Interventions: Behavioral: High Protein and Low Glycemic Index Diet
- Conventional Diet (Active Comparator): A protocol of a conventional diet.
  Interventions: Behavioral: Conventional Diet

INTERVENTIONS:
Behavioral: High Protein and Low Glycemic Index Diet — It will be evaluated a type of high protein diet with 1,3g/kg/day in kidney transplant recipients over 1 year after transplantation.
  Arms: High Protein and Low Glycemic Index Diet
Behavioral: Conventional Diet — Conventional diet over 1 year after transplantation.
  Arms: Conventional Diet

SUMMARY:
This study is a randomized clinical trial, which will follow and evaluate 120 kidney transplant recipients over one year. There will be two groups: a control group and the intervention group. The dietitian visits will happen monthly during the first six months and twice in the last six months.The intervention group will receive a high-protein and low glycemic index diet (1,3g/kg/day of protein) and the control group will keep following the hospital standard protocol. The study assessments (weight, anthropometry and biochemistry) will be performed during these visits over one year after the randomization period.

DETAILED DESCRIPTION:
Kidney transplantation is the greater renal replacement therapy and, compared with dialysis,is associated with better quality of life and reduced costs over time. However, it is well known that significant weight gain and obesity are very common after kidney transplantation, mainly during the first year after transplant. Besides, obesity is a risk factor for the development of cardiovascular complications, new-onset diabetes after transplantation and it is associated with graft loss. The use of immunosuppressive medications, the break of dietary restrictions associated with dialysis period and improvements in appetite are acceptable causes for weight gain. However, there is a lack of evidence for effective nutritional interventions to prevent weight gain after kidney transplant.

In this context, it is well known that high-protein and low glycemic index diets are effective for body weight loss and subsequent weight maintenance. Moreover, protein generally exerts a better satiety effect than carbohydrates and lipids. So that, considering that there is a need to develop effective interventions to minimize the negative impact of weight gain and obesity on kidney transplant outcomes, a randomized clinical trial, that evaluate the effect of a high protein and low glycemic index diet (as a nutritional intervention) is likely to be effective in preventing weight gain after kidney transplantation.

This study is a randomized clinical trial, which will follow and evaluate kidney transplant recipients during one year after transplantation. There will be two groups: a control group (60 patients) and the intervention group (60 patients). The dietitian visits will happen monthly at the first six months and twice in the last six months. The study assessments (weight, anthropometry, body composition and biochemistry) will be performed during these visits. Potential participants will be identified during their initial two months following transplantation. Eligible transplant recipients will be invited to participate, given detailed information about the trial and, if agreeable, will be asked to provide written informed consent. Participants will be randomized to receive either nutrition intervention with a high-protein and low glycemic index diet or an standard nutrition protocol. This randomization will be performed by a statistical consultant using randomization.com site. The length of the study will be 1 year for each patient, so that the assessment of anthropometry, including measures of weight (monthly) and body composition (every three months) will be performed by one specialist renal dietitian. Laboratory staff will perform all laboratories testing, including serum and urine creatinine (monthly), glycemia, cholesterol, HDL-cholesterol, triglycerides, glycated hemoglobin and uric acid (each three months), high-sensitivity C- reactive protein (baseline and 6th month) and 24-h urine test with albumin, protein, creatinine and urea excretion (every three months for intervention group and at baseline, 3rd, 6th and 12th month for control group). Demographic and clinical data will be assessed at the first dietitian visit. Body weight and height of patients will be obtained and body mass index (BMI) (kg/m2) will be calculated. Waist circumference will be measured midway between the lowest rib margin and the iliac crest, with flexible, nonstretched fiberglass tape. This evaluation will be made every visit (monthly in the first 6 months and twice in the last 6 months). Body fat percentage (assessed each three months) will be measured by using tetrapolar bioimpedance and basal metabolic rate will be evaluated by indirect calorimetry at baseline and 6 months later. All the anthropometric assessment will be performed with the patient fasting, wearing light clothing, without contact with metals and without shoes. The prescription of the diet will be calculated by using nutritional table by software version. It will be considered 1,3g /kg/day of protein and the glycemic index will be estimated with glucose as standard food. Energy intake will be assessed by a 24-h recall on the day of each dietitian visit by the research dietitian. Diet composition also will be analyzed by using nutritional table by software and will be made in every visit. Satiety levels will be assessed each three months for intervention group and only at baseline for control group by using a visual analogue scale of appetite.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients

Exclusion Criteria:

* Younger than 18
* Prior Transplant
* Multiple organ transplant
* Cancer
* Women in pregnancy or lactation period
* Recipients of living donors
* Urinary albumin excretion> 300 mg / 24h.
* Glomerular filtration rate <30 mL / min / 1.73

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Weight Change | Baseline, 1st month, 2nd month, 3rd month, 4th month, 5th month, 6th month, 9th month and 12th month.
  Digital Balance

SECONDARY OUTCOMES:
Body Composition Change | Baseline, 3rd month, 6th month, 9th month and 12th month.
  Bioelectrical impedance analysis
Basal Metabolic Rate | Baseline and 6th month.
  Indirect Calorimetry
Satiety | Baseline, 3rd month, 6th month, 9th month and 12th month for intervention group and at baseline for control group.
  Visual analogue scale of appetite
Kidney function | 12 months
  Kidney function will be assessed monthly over one year through serum creatinine with estimated glomerular filtration rate by Modification of Diet in Renal Disease equation.
Glycated hemoglobin | Baseline, 3rd month, 6th month, 9th month and 12th month.
  Glycated hemoglobin Laboratory Test
Lipid Profile | Baseline, 3rd month, 6th month, 9th month and 12th month.
  Total cholesterol level
Inflammation | Baseline and 6th month.
  High-Sensitivity C-Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Elis Forcellini Pedrollo, Master, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedrollo EF, Correa C, Nicoletto BB, de Melo Cardoso de Freitas J, Buboltz JR, da Costa BDF, Dos Santos Guedes G, Bauer AC, Manfro RC, Souza GC, Leitao CB. Effect of an intensive nutrition intervention of a high protein and low glycemic load diet on weight of kidney transplant recipients: a randomized clinical trial. Endocrine. 2025 Jan;87(1):106-115. doi: 10.1007/s12020-024-03978-y. Epub 2024 Aug 5. PMID 39102111
- [Derived] Pedrollo EF, Nicoletto BB, Carpes LS, de Freitas JMC, Buboltz JR, Forte CC, Bauer AC, Manfro RC, Souza GC, Leitao CB. Effect of an intensive nutrition intervention of a high protein and low glycemic-index diet on weight of kidney transplant recipients: study protocol for a randomized clinical trial. Trials. 2017 Sep 6;18(1):413. doi: 10.1186/s13063-017-2158-2. PMID 28874181